CLINICAL TRIAL: NCT07026422
Title: Iparomlimab/Tuvonralimab Integrating With Total Neoadjuvant Therapy for pMMR/MSS Locally Advanced Rectal Cancer (IT-TNT): A Single-arm, Exploratory, Phase II Trial
Brief Title: Iparomlimab/Tuvonralimab Integrating With Total Neoadjuvant Therapy for pMMR/MSS Locally Advanced Rectal Cancer (IT-TNT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Radiation Oncology Department, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-151-02
Record Dates: First submitted 2025-05-21; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Rectal Malignant Neoplasms
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual immunotherapy group (Experimental): Total neoadjuvant therapy integrating iparomlimab/tuvonralimab with chemoradiotherapy
  Interventions: Combination Product: Total neoadjuvant therapy integrating iparomlimab/tuvonralimab with chemoradiotherapy

INTERVENTIONS:
Combination Product: Total neoadjuvant therapy integrating iparomlimab/tuvonralimab with chemoradiotherapy — 1. Radiotherapy:
     Radiotherapy location: primary site and the corresponding draining lymph node. Radiotherapy techniques: IMRT/VMRT.
     Radiotherapy dose and fractionation pattern: conventional external irradiation, 50Gy/25 fx/5 weeks or 25Gy/5fx/1 week.
  2. Chemotherapy:
  Long-course radiotherapy concurrent with chemotherapy: capecitabine 825mg/m2, bid, d1-5/week.
  Short-course radiotherapy without concurrent chemotherapy. Consolidation chemotherapy and immunotherapy: QL1706 (iparomlimab and tuvonralimab 5mg/kg, d1) and CAPOX (Oxaliplatin 130mg/m2, d1 + capecitabine 1000mg/m2, bid, d1-14), repeated on a 21-day cycle, for 6 cycles. 3. Surgery or watch-and-wait Total mesorectal excision (TME), or watch-and-wait (for patients with clinical complete response).

SUMMARY:
In colorectal cancer (CRC), ICIs show strong therapeutic associations with microsatellite instability-high (MSI-H) status, while patients with proficient mismatch repair/microsatellite stable (pMMR/MSS) tumors exhibit poor responses. Dual immunotherapy may represent a promising strategy for MSS populations. The Dutch NICHE trial reported a 27% pathological response rate (4/15) in MSS CRC patients with clinical stage I-III disease treated with neoadjuvant ipilimumab plus nivolumab. In advanced or metastatic CRC, a study by Jin Li et al. demonstrated that iparomlimab/tuvonralimab combined with bevacizumab and the XELOX regimen achieved an objective response rate of 70.6% (95% CI: 56.2%-82.5%).

Radiotherapy may synergize with ICIs through multiple immunomodulatory mechanisms. For pMMR/MSS LARC, combining CRT with ICIs holds promise to overcome the "immune-cold" tumor microenvironment and improve therapeutic efficacy. In this clinical trial, the investigators aim to evaluate the efficacy and safety of integrating immunotherapy with CRT as a novel total neoadjuvant therapy for pMMR/MSS rectal cancer.

DETAILED DESCRIPTION:
The "sandwich" approach, combining preoperative concurrent chemoradiotherapy (CRT) with total mesorectal excision (TME) and postoperative adjuvant chemotherapy, has been shown to improve pathological complete response (pCR) rates, local control rates (LCR), and sphincter preservation rates in patients with locally advanced rectal cancer (LARC). However, this strategy does not significantly enhance overall survival (OS) or distant metastasis-free survival (DMFS). Total neoadjuvant therapy (TNT), a novel treatment paradigm, involves administering chemotherapy either before neoadjuvant CRT (induction TNT) or after neoadjuvant CRT (consolidation TNT). This approach improves treatment compliance, reduces chemotherapy-related toxicity, and increases pCR rates. Patients achieving pCR following TNT exhibit lower risks of local tumor recurrence and improved survival outcomes.

Immune checkpoint inhibitors (ICIs) have become a cornerstone of cancer therapy. Antibodies targeting negative immune regulators-such as cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), programmed cell death-1 (PD-1), and programmed cell death ligand 1 (PD-L1)-have demonstrated efficacy across multiple solid tumors. In colorectal cancer (CRC), ICIs show strong therapeutic associations with microsatellite instability-high (MSI-H) status, while patients with proficient mismatch repair/microsatellite stable (pMMR/MSS) tumors exhibit poor responses. Dual immunotherapy may represent a promising strategy for MSS populations. The Dutch NICHE trial reported a 27% pathological response rate (4/15) in MSS CRC patients with clinical stage I-III disease treated with neoadjuvant ipilimumab (anti-CTLA-4) plus nivolumab (anti-PD-1), including 3 major pathological responses and 1 partial response. In advanced or metastatic CRC, a study by Jin Li et al. demonstrated that iparomlimab/tuvonralimab combined with bevacizumab and the XELOX regimen achieved an objective response rate of 70.6% (95% CI: 56.2%-82.5%).

Radiotherapy may synergize with ICIs through multiple immunomodulatory mechanisms, including enhanced tumor antigen release, activation of innate immune pathways, increased T-cell infiltration, improved antigen presentation, and modulation of immunosuppressive cells. For pMMR/MSS LARC, combining CRT with ICIs holds promise to overcome the "immune-cold" tumor microenvironment and improve therapeutic efficacy. In this clinical trial, the investigators aim to evaluate the efficacy and safety of integrating immunotherapy with CRT as a novel total neoadjuvant therapy for pMMR/MSS rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, male and female
2. Histologically confirmed pMMR/MSS rectal adenocarcinoma, defined by MRI as clinical stage II (T3-4, N-) or stage III (any T, N+)
3. Tumor within 12 cm of the anal verge with at least one of the following high-risk factors: cT4, cN2, extramural vascular invasion [EMVI+], mesorectal fascia involved [MRF+], lateral lymph node [LN+], tumor deposit, or low rectal cancer (≤5 cm from the anal verge)
4. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
5. No evidence of distant metastases based on chest and abdominal CT or whole body PET-CT examinations
6. No other rectal cancer (e.g., sarcoma, lymphoma, carcinoid, squamous cell carcinoma, neuroendocrine carcinoma, etc.) or synchronous colon cancer
7. Presence of measurable lesions that meet RECIST v1.1 criteria for evaluation.

Exclusion Criteria:

1. dMMR or MSI-H patients
2. Myelosuppression without obvious causes
3. Locally advanced rectal cancer without high-risk factors
4. Prior or concurrent other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix)
5. Severe allergic reaction to other monoclonal antibodies
6. Uncontrolled cardiac clinical symptoms or disease
7. Active autoimmune disease or immunodefciencies, known history of organ transplantation or systematic use of immunosuppressive agents
8. Abnormal coagulation (INR>1.5 or PT>16s), bleeding tendency or on thrombolytic or anticoagulant therapy
9. Known history and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonitis, or severely impaired lung function
10. Known history of prior antitumor therapy, including radiotherapy, chemotherapy, immune checkpoint inhibitors, T-cell related therapy, etc.
11. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1-2 antibody-positive), active syphilis infection, active tuberculosis infection, or active hepatitis B virus or hepatitis C virus infection at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall complete response (CR) rate | 1 year
  Overall complete response (CR) rate, meaning the rates of pathological complete response (pCR) plus clinical complete response (cCR).

SECONDARY OUTCOMES:
Overall survival (OS) | 3 year
  From date of radiotherapy initiation until the date of death from any cause or last follow-up, whichever came first.
Rate of surgical complications | 1 year
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.
Organ preservation rate | 1 year
3 year disease free survival (DFS) rate | 3 year
  From date of surgery completion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
3 year local recurrence free survival (LRFS) rate | 3 year
  Time Frame: From date of surgery completion until the date of first documented pelvic failure, assessed up to 36 months
The incidence and grade of adverse events | 1 year
  The incidence and grade of adverse events, determined according to NCI-CTCAE 5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Docter, Principal Investigator — Shandong Cancer Hospital and Institute, Department of Radiation Oncology
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No